CLINICAL TRIAL: NCT00136630
Title: Natural History, Genetic Bases and Phenotype-genotype Correlations in Autosomal Dominant Spinocerebellar Degenerations
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: RBM01-59 _ AOM03059
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Spinocerebellar Ataxias; Spastic Paraplegias
Keywords: dominant spinocerebellar degenerations; new rate scales; natural history; molecular biology; candidate genes
MeSH Terms: conditions — Spinocerebellar Ataxias; Paraplegia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective

SUMMARY:
The autosomal dominant spinocerebellar degenerations are a highly heterogeneous, clinically and genetically, group of rare diseases and of severe evolution. So far, the responsible genes for less than 50% of the cases are known and because of their rarity, there are no phenotype-genotype correlations and well-defined disease history.

The aims of the project are to develop and validate quantitative tools of the cerebellar syndrome and of the spasticity, to establish links between the phenotype and the result of the molecular analysis, to identify new loci/genes responsible for these disorders, and to establish the natural history of the disease according to the genotype.

To this end, a prospective and multicentric study is proposed for recruiting and evaluating, clinically, a cohort of 225 patients; 150 of them are already followed-up in the centers involved. A DNA collection will be set up in order to search for the implication of new loci and genes. A clinico-genetic database will be set up combining data from successive clinical evaluations and those of genotyping.

This strategy will allow access to genetic counselling and molecular diagnosis (positive, presymptomatic or prenatal diagnoses), based on a rational strategy from phenotype-genotype correlations and the information concerning the relative frequency of the genes. The detailed description, with the help of new evaluation tools and of the follow-up of the natural history of the disease according to the genotype, constitutes a crucial step in the design of therapeutical trials in these orphan disorders. Furthermore, the regular follow-up by specialized centers will allow better care of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Progressive ataxia or paraplegia,
* Familial history of the disease (patients),
* Over 18 years of age
* No presentation of neurological or osteoarticular disorders

Exclusion Criteria:

* Refusal to participate in the protocol,
* An unknown familial history,
* Presenting with an interrecurrent disorder making the evaluation of the disease (stroke, dementia) impossible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: French population
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2005-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Dürr, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Broussolle Emmanuel, MD, PhD, Principal Investigator — Hôpitaux Civils de Lyon; Pierre Labauge, MD, PhD, Principal Investigator — Hôpitaux de Nîmes; Cyril Goizet, MD, Principal Investigator — Hôpitaux de Bordeaux; Patrick Calvas, MD, PhD, Principal Investigator — Hôpitaux de Toulouse; Jean-Philippe Azulay, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Marseille; Didier Hannequin, MD, PhD, Principal Investigator — Hôpitaux de Rouen; Pierre Pollak, MD, PhD, Principal Investigator — Hôpitaux de Grenoble
Locations (8):
- France (8):
  - Hôpital Pellegrin, Bordeaux
  - CHU de Grenoble, Grenoble
  - Hôpital Neurologique Pierre Wertheimer, Lyon
  - Hôpital La Timone, Marseille
  - Hôpital Carémeau, Nîmes
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Purpan, Toulouse

REFERENCES:
- [Result] Klebe S, Durr A, Rentschler A, Hahn-Barma V, Abele M, Bouslam N, Schols L, Jedynak P, Forlani S, Denis E, Dussert C, Agid Y, Bauer P, Globas C, Wullner U, Brice A, Riess O, Stevanin G. New mutations in protein kinase Cgamma associated with spinocerebellar ataxia type 14. Ann Neurol. 2005 Nov;58(5):720-9. doi: 10.1002/ana.20628. PMID 16193476
- [Result] Stevanin G, Hahn V, Lohmann E, Bouslam N, Gouttard M, Soumphonphakdy C, Welter ML, Ollagnon-Roman E, Lemainque A, Ruberg M, Brice A, Durr A. Mutation in the catalytic domain of protein kinase C gamma and extension of the phenotype associated with spinocerebellar ataxia type 14. Arch Neurol. 2004 Aug;61(8):1242-8. doi: 10.1001/archneur.61.8.1242. PMID 15313841
- [Result] Stevanin G, Durr A, Dussert C, Penet C, Brice A. Mutations in the FGF14 gene are not a major cause of spinocerebellar ataxia in Caucasians. Neurology. 2004 Sep 14;63(5):936. doi: 10.1212/01.wnl.0000137020.30604.1e. No abstract available. PMID 15365159
- [Result] Waters MF, Minassian NA, Stevanin G, Figueroa KP, Bannister JP, Nolte D, Mock AF, Evidente VG, Fee DB, Muller U, Durr A, Brice A, Papazian DM, Pulst SM. Mutations in voltage-gated potassium channel KCNC3 cause degenerative and developmental central nervous system phenotypes. Nat Genet. 2006 Apr;38(4):447-51. doi: 10.1038/ng1758. Epub 2006 Feb 26. PMID 16501573
- [Result] Depienne C, Tallaksen C, Lephay JY, Bricka B, Poea-Guyon S, Fontaine B, Labauge P, Brice A, Durr A. Spastin mutations are frequent in sporadic spastic paraparesis and their spectrum is different from that observed in familial cases. J Med Genet. 2006 Mar;43(3):259-65. doi: 10.1136/jmg.2005.035311. Epub 2005 Jul 31. PMID 16055926
- [Result] Depienne C, Fedirko E, Forlani S, Cazeneuve C, Ribai P, Feki I, Tallaksen C, Nguyen K, Stankoff B, Ruberg M, Stevanin G, Durr A, Brice A. Exon deletions of SPG4 are a frequent cause of hereditary spastic paraplegia. J Med Genet. 2007 Apr;44(4):281-4. doi: 10.1136/jmg.2006.046425. Epub 2006 Nov 10. PMID 17098887
- [Result] Depienne C, Fedirko E, Faucheux JM, Forlani S, Bricka B, Goizet C, Lesourd S, Stevanin G, Ruberg M, Durr A, Brice A. A de novo SPAST mutation leading to somatic mosaicism is associated with a later age at onset in HSP. Neurogenetics. 2007 Aug;8(3):231-3. doi: 10.1007/s10048-007-0090-4. Epub 2007 Jun 28. PMID 17597328
- [Result] Hanein S, Durr A, Ribai P, Forlani S, Leutenegger AL, Nelson I, Babron MC, Elleuch N, Depienne C, Charon C, Brice A, Stevanin G. A novel locus for autosomal dominant "uncomplicated" hereditary spastic paraplegia maps to chromosome 8p21.1-q13.3. Hum Genet. 2007 Nov;122(3-4):261-73. doi: 10.1007/s00439-007-0396-1. Epub 2007 Jun 28. PMID 17605047
- [Result] Ribai P, Depienne C, Fedirko E, Jothy AC, Viveweger C, Hahn-Barma V, Brice A, Durr A. Mental deficiency in three families with SPG4 spastic paraplegia. Eur J Hum Genet. 2008 Jan;16(1):97-104. doi: 10.1038/sj.ejhg.5201922. Epub 2007 Oct 24. PMID 17957230
- [Result] du Montcel ST, Charles P, Ribai P, Goizet C, Le Bayon A, Labauge P, Guyant-Marechal L, Forlani S, Jauffret C, Vandenberghe N, N'guyen K, Le Ber I, Devos D, Vincitorio CM, Manto MU, Tison F, Hannequin D, Ruberg M, Brice A, Durr A. Composite cerebellar functional severity score: validation of a quantitative score of cerebellar impairment. Brain. 2008 May;131(Pt 5):1352-61. doi: 10.1093/brain/awn059. Epub 2008 Mar 31. PMID 18378516
- [Result] Goizet C, Boukhris A, Mundwiller E, Tallaksen C, Forlani S, Toutain A, Carriere N, Paquis V, Depienne C, Durr A, Stevanin G, Brice A. Complicated forms of autosomal dominant hereditary spastic paraplegia are frequent in SPG10. Hum Mutat. 2009 Feb;30(2):E376-85. doi: 10.1002/humu.20920. PMID 18853458
- [Derived] Tezenas du Montcel S, Durr A, Rakowicz M, Nanetti L, Charles P, Sulek A, Mariotti C, Rola R, Schols L, Bauer P, Dufaure-Gare I, Jacobi H, Forlani S, Schmitz-Hubsch T, Filla A, Timmann D, van de Warrenburg BP, Marelli C, Kang JS, Giunti P, Cook A, Baliko L, Melegh B, Boesch S, Szymanski S, Berciano J, Infante J, Buerk K, Masciullo M, Di Fabio R, Depondt C, Ratka S, Stevanin G, Klockgether T, Brice A, Golmard JL. Prediction of the age at onset in spinocerebellar ataxia type 1, 2, 3 and 6. J Med Genet. 2014 Jul;51(7):479-86. doi: 10.1136/jmedgenet-2013-102200. Epub 2014 Apr 29. PMID 24780882
- [Derived] Tezenas du Montcel S, Charles P, Goizet C, Marelli C, Ribai P, Vincitorio C, Anheim M, Guyant-Marechal L, Le Bayon A, Vandenberghe N, Tchikviladze M, Devos D, Le Ber I, N'Guyen K, Cazeneuve C, Tallaksen C, Brice A, Durr A. Factors influencing disease progression in autosomal dominant cerebellar ataxia and spastic paraplegia. Arch Neurol. 2012 Apr;69(4):500-8. doi: 10.1001/archneurol.2011.2713. PMID 22491195
- See also: Related Info — http://www.aphp.fr